CLINICAL TRIAL: NCT03604029
Title: Evaluating the Diagnostic Performance of Near Infrared Spectroscopy (NIRS) in the Setting of Acute Compartment Syndrome (ACS) in Traumatized Lower Extremities
Brief Title: Evaluating the Diagnostic Performance of ACS Using NIRS in Traumatized Lower Extremities
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: W81XWH17C0029
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Compartment Syndrome of Leg
Keywords: ACS
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Qualifying Subjects: Qualifying subjects who are high risk for ACS.
  Interventions: Device: Near Infrared Spectroscopy
- Qualifying Subjects with ACS: Qualifying subjects who are diagnosed with ACS
  Interventions: Device: Near Infrared Spectroscopy

INTERVENTIONS:
Device: Near Infrared Spectroscopy — Near Infrared Spectroscopy (NIRS) sensors are applied to injured leg compartments and a control compartment to continuously measure tissue oxygenation.

SUMMARY:
This is a study intended to validate a new set of guidelines for a device that uses light to measure the amount of oxygen in the muscles of injured and non-injured legs and forearms in specific situations.

DETAILED DESCRIPTION:
This is a study intended to validate a new set of guidelines for a device that uses light to measure the amount of oxygen in the muscles of injured and non-injured legs and forearms in specific situations. The name of this technology is NIRS (near-infrared spectroscopy). We have shown NIRS can be helpful in diagnosing ACS. We think two of the primary advantages of this device are that it is noninvasive (not painful) and it collects data continuously, so that if the disease develops, it can be detected early and treated appropriately. We have studied the capabilities of NIRS for many years. The last step in the process of proving NIRS and its use in ACS will be to test our recommendations and guidelines. The goal of this study is to test and prove our clinical guidelines we developed through previous work. This is an interventional study, which means the data we collect will be used to manage the patient and their care.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years
2. Ability to be enrolled within 12 hours of qualifying injury
3. Must have at least one uninjured upper or lower extremity
4. Must have a "severe leg injury" meeting one of the following anatomical locations and mechanisms of injury.

Anatomic Location:

1. Tibia/fibula shaft fracture
2. Tibial plateau fracture (including lateral split depression, lateral depression, medial plateau, bicondylar, and bicondylar with metaphyseal extension)
3. Gunshot wound to leg without tibia fracture

High Energy Mechanism of Injury (MOI):

1. Fall from more than 5-foot height
2. Motor vehicle collision (more than 15mph)
3. Motor vehicle versus pedestrian accident
4. High velocity gunshot wound (with or without tibia fracture)
5. Crush injury
6. Sport/recreation

Exclusion Criteria:

1. Application of NIRS monitoring would be an impediment to care
2. Known prior injury, surgery, or disease of the lower extremity (including thigh) that alters normal circulation in the leg (including peripheral vascular disease)
3. Admission for atraumatic medical reasons (i.e. myocardial infarction, sepsis)
4. Consent cannot be obtained from the patient or their LAR within 12 hours of injury
5. Has already undergone fasciotomy of the injured leg prior to enrollment
6. Has spinal injuries that result in complete loss of function (complete spinal cord injuries)
7. Has bilateral upper and lower extremity injuries greater than simple soft tissue injuries
8. Is in police custody at presentation to the hospital
9. Is a woman who is pregnant
10. Has open injury on the injured leg that is large enough that at least two NIRS sensor cannot be safely placed. At a minimum two sensors must be placed on the injured leg(s).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the trauma bay, surgical wards and ICU of the four participating facilities. This study will enroll approximately 300 subjects over four sites: Piedmont Athens Regional Medical Center, Grady Memorial Hospital, Mayo Clinic, and San Antonio Military Medical Center, over a period of approximately 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute Compartment Syndrome | Zero to seventy two hours from enrollment.
  The subject develops and diagnosed with Acute Compartment Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Chevas R. Yeoman, MPH, Study Director — The Geneva Foundation; William M. Reisman, MD, Principal Investigator — Emory Department of Orthopedics; Charles L. Ogburn, MD, Principal Investigator — Athens Orthopedic Clinic; Patrick M. Osborn, MD, Principal Investigator — San Anontio Military Medical Center; Brandon J. Yuan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Brett A. Freedman, Col, MD, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available to other researchers.

REFERENCES:
- [Result] Reisman WM, Shuler MS, Roskosky M, Kinsey TL, Freedman BA. Use of Near-Infrared Spectroscopy to Detect Sustained Hyperaemia Following Lower Extremity Trauma. Mil Med. 2016 Feb;181(2):111-5. doi: 10.7205/MILMED-D-14-00689. PMID 26837078
- [Result] Shuler MS, Roskosky M, Kinsey T, Glaser D, Reisman W, Ogburn C, Yeoman C, Wanderman NR, Freedman B. Continual near-infrared spectroscopy monitoring in the injured lower limb and acute compartment syndrome: an FDA-IDE trial. Bone Joint J. 2018 Jun 1;100-B(6):787-797. doi: 10.1302/0301-620X.100B6.BJJ-2017-0736.R3. PMID 29855235